CLINICAL TRIAL: NCT05408936
Title: Study of the Mechanisms Leading to Increased Hemoglobin Levels and of the Cardiorenal Response in Type 2 Diabetic Patients With Recent Initiation of SGLT2 Inhibitors.
Brief Title: SGLT2 Inhibitors and Effects on Hematopoiesis, Inflammation and Metabolic Markers
Acronym: SGLT2HgB
Status: Active, not recruiting | Type: Observational
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Ioannis Habeos, Professor, University of Patras
Other Study IDs: 59/15.02.2022
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: SGLT2 inhibitors, hemoglobin, NTproBNP, ketones
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Ketosis | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, urine
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: SGLT2 inhibitor — Patients receive an SGLT2 inhibitor as part of theirn routine care.

SUMMARY:
Study of the response to SGLT2 inhibitors in type 2 diabetic patients with relevance to the erythropoesis and indexes of cardiorenal function.

The study enrolls type 2 diabetic patients in whom the introduction of a SGLT2 inhibitor is deemed necessary as part of their routine treatment during their visit to our outpatient diabetes unit.

A whole blood, a serum and a urine sample is obtained before and one month after the initiation of treatment with a SGLT2 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* Hba1C>7% on their current treatment
* introduction of SGLT2 inhibitor as part of their routine care

Exclusion Criteria:

* eGFR<60 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients who visit the diabetes outpatient clinic in the University Hospital of Patras, Greece
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | 0-1-3 months
Erythropoetin | 0-1-3 months
NT-proBNP | 0-1-3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Patras, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Data available upon reasonable request